CLINICAL TRIAL: NCT03444103
Title: Safety, Tolerability and Efficacy of Anti-IL-6 Antibody Clazakizumab in Late Antibody-Mediated Rejection After Kidney Transplantation - a Pilot Trial
Brief Title: A Pilot Trial of Clazakizumab in Late ABMR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: CSL Behring (Industry); University of Alberta (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Farsad Eskandary, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK1428/2017; 2017-001604-30 (EudraCT Number)
Record Dates: First submitted 2018-01-16; First posted 2018-02-23 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Antibody-mediated Rejection
Keywords: IL-6 blockade
MeSH Terms: interventions — clazakizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clazakizumab / Clazakizumab (Active Comparator): Monthly subcutaneous injections of 25mg clazakizumab for three months (after completion of part A, monthly injection of 25mg clazakizumab for nine months).
  Interventions: Drug: Clazakizumab / Clazakizumab
- Placebo / Clazakizumab (Placebo Comparator): Monthly subcutaneous injections of placebo (saline) for three months (after completion of part A, monthly injection of 25mg clazakizumab for nine months).
  Interventions: Drug: Placebo / Clazakizumab

INTERVENTIONS:
Drug: Clazakizumab / Clazakizumab — Humanized monoclonal anti-IL-6 antibody
  Other Names: Anti-IL-6 antibody
  Arms: Clazakizumab / Clazakizumab
Drug: Placebo / Clazakizumab — 0.9% Saline
  Other Names: Saline
  Arms: Placebo / Clazakizumab

SUMMARY:
This bi-center study (Medical University of Vienna & Charité Berlin) is an investigator-driven pilot trial designed to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy (preliminary assessment) of humanized anti-IL-6 monoclonal antibody clazakizumab in kidney transplant recipients with late antibody-mediated rejection (ABMR). The study is designed as a phase 2 trial and has two subsequent sub-parts, a randomized placebo-controlled trial (part A) of 12 weeks, where recipients are allocated to receive either anti-IL-6 antibody clazakizumab (n=10) or placebo (n=10), followed by an open-label prospective study, where all 20 study patients will receive clazakizumab for a period of 40 weeks. Study protocol biopsies will be performed at the end of part A and part B.

DETAILED DESCRIPTION:
Part A:

Patients positive for anti-HLA donor-specific antibodies (DSA) and with biopsy-proven late ABMR (Acute/active or chronic/active phenotype according to the Banff 2015 classification) will be identified and recruited at the kidney transplantation outpatient services of the two center sites. Participants will be randomized to receive either clazakizumab or placebo subcutaneously (1:1 randomization stratified for ABMR type) for a period of 12 weeks (administration of clazakizumab/placebo at day 0, and after 4 and 8 weeks). After 12 weeks, patients will be subjected to a first follow-up biopsy. Primary goals of this part of the trial are to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of a short course of treatment. Moreover, part A will allow for a first preliminary assessment of the impact of clazakizumab on ABMR-associated inflammation detected in peripheral blood and in the rejecting organ allograft, on the pharmacokinetics of pantoprazole as a probe drug to investigate influence of IL-6 blockade on cytochrome P450 (CYP) dependent drug metabolism (potential effects on the half-life of CYP-metabolized drugs such as pantoprazole, and on the short-term course of DSA mean fluorescence intensity (MFI) and kidney allograft function (eGFR, urinary protein excretion). The randomization sequence will be unblinded for a first data analysis after the last patient has completed the 12-week follow-up period.

Part B:

After completion of part A after 12 weeks, all study patients will enter part B, an open-label part of the study. All 20 subjects will receive subcutaneous clazakizumab in 4-weekly intervals until the end-of-study (EOS) visit after 52 weeks and will then be subjected to a second protocol biopsy. Major goals of part B are to evaluate the safety and tolerability of a prolonged period of treatment with clazakizumab and the long-term impact of this antibody on the evolution of ABMR, rejection-associated biomarkers and kidney allograft function and survival over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Age >18 years
* Functioning living or deceased donor allograft after ≥365 days post-transplantation
* eGFR >30 ml/min/1.73 m2
* Detection of HLA class I and/or II antigen-specific antibodies (preformed and/or de novo DSA).
* Acute/active or chronic/active ABMR (±C4d in PTC) according to Banff 2013/2015
* Molecular ABMR score (ABMRpm) ≥0.2

Exclusion Criteria:

* Patients actively participating in another clinical trial
* Age ≤18 years
* Female subject is pregnant or lactating
* Index biopsy results:
* T-cell-mediated rejection classified Banff grade ≥I
* De novo or recurrent severe thrombotic microangiopathy
* Polyoma virus nephropathy
* De novo or recurrent glomerulonephritis
* Acute rejection treatment <3 month before screening
* Acute deterioration of graft function (eGFR decline within 1-3 months >25%)
* Nephrotic range proteinuria >3500 mg/g protein/creatinine ratio
* Active viral, bacterial or fungal infection precluding intensified immunosuppression
* Active malignant disease precluding intensified immunosuppressive therapy
* Abnormal liver function tests (ALT, AST, bilirubin > 1.5 x upper limit of normal)
* Other significant liver disease
* Latent or active tuberculosis (positive QuantiFERON-TB-Gold test, Chest X-ray)
* Administration of a live vaccine within 6 weeks of screening
* Neutropenia (<1 G/L) or thrombocytopenia (<100 G/L)
* History of gastrointestinal perforation, diverticulitis, or inflammatory bowel disease
* Allergy against proton pump inhibitors
* History of alcohol or illicit substance abuse
* Serious medical or psychiatric illness likely to interfere with participation in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and severe adverse events (AE's, SAE's) | 12 months
  Serious and Non-Serious adverse events probably or possibly attributable to clazakizumab

SECONDARY OUTCOMES:
Anti-clazakizumab antibodies in serum | At 0, 12 and 52 weeks
  - Concentration of anti-clazakizumab antibodies in serum (ng/mL)
Clazakizumab serum concentration | At 0, 12 and 52 weeks
  - Total clazakizumab serum concentration (ng/mL)
Pantoprazole serum concentration | At 0, 12 and 52 weeks
  - Effect of clazakizumab on pantoprazole serum concentration (nanogram per mL)
Protocol biopsy results - microcirculation inflammation | At week 11 and at week 52
  - Microcirculation inflammation (g+ptc score), scale 0-3, higher = worse prognosis
Protocol biopsy results - chronic damage | At week 11 and at week 52
  - Transplant glomerulopathy (cg) and interstitial fibrosis/tubular atrophy (IFTA) scores, scale 0-3, higher = worse prognosis
Protocol biopsy results - molecular signs of ABMR | At week 11 and at week 52
  - Molecular ABMR score (molecular microscope, MMDx), scale 0-1 in 0.1 steps, higher = worse prognosis
Protocol biopsy results - ABMR phenotype | At week 11 and at week 52
  - Archetype analysis of gene expression profiles (molecular microscope, MMDx), ABMR archetype score, scale 0-1 in 0.1 steps, higher = worse prognosis
Anti-HLA antibody levels - antibody strength | At 0, 12 and 52 weeks
  - Maximum and sum of mean fluorescence intensity (MFI) of DSA (Luminex) - higher is worse
Anti-HLA antibody levels - number of DSA | At 0, 12 and 52 weeks
  - Number of DSA (Luminex) - more is worse
Anti-HLA antibody levels - broadness of antibody reactivity | At 0, 12 and 52 weeks
  - Broadness of sensitization (virtual PRA, Luminex), scale: %, higher = worse
Allograft function - eGFR | At day 0, week 1, 2, 3, 4, 5, 6, 7, 8, 11, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 51 and 52
  - Estimated GFR (CKD-EPI, mL/min/1.73m2)
Allograft function - protein excretion in spot urine | At day 0, week 1, 2, 3, 4, 5, 6, 7, 8, 11, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 51 and 52
  - Urinary protein excretion in spot urine (protein/creatinine ratio in mg/g)
Total IgG concentration | At 0, 12 and 52 weeks
  - Nephelometry, mg/dL
Total IgM concentration | At 0, 12 and 52 weeks
  - Nephelometry, mg/dL
Total IgA concentration | At 0, 12 and 52 weeks
  - Nephelometry, mg/dL
IgG subclass 1 (IgG1) | At 0, 12 and 52 weeks
  - ELISA, mg/dL
IgG subclass 2 (IgG2) | At 0, 12 and 52 weeks
  - ELISA, mg/dL
IgG subclass 3 (IgG3) | At 0, 12 and 52 weeks
  - ELISA, mg/dL
IgG subclass 4 (IgG4) | At 0, 12 and 52 weeks
  - ELISA, mg/dL
Effect on leukocyte subsets in peripheral blood | At 0, 12 and 52 weeks
  - Fluorescence intensity (0 to no upper limit)
Cytokine patterns and endothelial activation/injury markers in serum | At 0, 12 and 52 weeks
  - Luminex bead panels, mean fluorescence intensities (MFI)
Effect on IL-6 gene expression in peripheral blood cells | At 0, 12 and 52 weeks
  rtPCR
Effect on IL-6R gene expression in peripheral blood cells | At 0, 12 and 52 weeks
  rtPCR
Patient survival | 12 months
  Death: number of events, time to event
Graft survival | 12 months
  Graft loss: number of events, time to event
Occurrence of biopsy-proven acute rejection necessitating rejection treatment | At week 52
  Number of anti-rejection treatments with a substance other than the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University Vienna
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Charité University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mease PJ, Gottlieb AB, Berman A, Drescher E, Xing J, Wong R, Banerjee S. The Efficacy and Safety of Clazakizumab, an Anti-Interleukin-6 Monoclonal Antibody, in a Phase IIb Study of Adults With Active Psoriatic Arthritis. Arthritis Rheumatol. 2016 Sep;68(9):2163-73. doi: 10.1002/art.39700. PMID 27059799
- [Background] Choi J, Aubert O, Vo A, Loupy A, Haas M, Puliyanda D, Kim I, Louie S, Kang A, Peng A, Kahwaji J, Reinsmoen N, Toyoda M, Jordan SC. Assessment of Tocilizumab (Anti-Interleukin-6 Receptor Monoclonal) as a Potential Treatment for Chronic Antibody-Mediated Rejection and Transplant Glomerulopathy in HLA-Sensitized Renal Allograft Recipients. Am J Transplant. 2017 Sep;17(9):2381-2389. doi: 10.1111/ajt.14228. Epub 2017 Mar 10. PMID 28199785
- [Background] Eskandary F, Regele H, Baumann L, Bond G, Kozakowski N, Wahrmann M, Hidalgo LG, Haslacher H, Kaltenecker CC, Aretin MB, Oberbauer R, Posch M, Staudenherz A, Handisurya A, Reeve J, Halloran PF, Bohmig GA. A Randomized Trial of Bortezomib in Late Antibody-Mediated Kidney Transplant Rejection. J Am Soc Nephrol. 2018 Feb;29(2):591-605. doi: 10.1681/ASN.2017070818. Epub 2017 Dec 14. PMID 29242250
- [Derived] Mayer KA, Doberer K, Halloran PF, Budde K, Haindl S, Muhlbacher J, Eskandary F, Viard T, Casas S, Jilma B, Bohmig GA. Anti-interleukin-6 Antibody Clazakizumab in Antibody-mediated Kidney Transplant Rejection: Effect on Donor-derived Cell-free DNA and C-X-C Motif Chemokine Ligand 10. Transplant Direct. 2022 Nov 10;8(12):e1406. doi: 10.1097/TXD.0000000000001406. eCollection 2022 Dec. PMID 36382130
- [Derived] Muhlbacher J, Schorgenhofer C, Doberer K, Durr M, Budde K, Eskandary F, Mayer KA, Schranz S, Ely S, Reiter B, Chong E, Adler SH, Jilma B, Bohmig GA. Anti-interleukin-6 antibody clazakizumab in late antibody-mediated kidney transplant rejection: effect on cytochrome P450 drug metabolism. Transpl Int. 2021 Aug;34(8):1542-1552. doi: 10.1111/tri.13954. Epub 2021 Jul 8. PMID 34153143
- [Derived] Eskandary F, Durr M, Budde K, Doberer K, Reindl-Schwaighofer R, Waiser J, Wahrmann M, Regele H, Spittler A, Lachmann N, Firbas C, Muhlbacher J, Bond G, Halloran PF, Chong E, Jilma B, Bohmig GA. Clazakizumab in late antibody-mediated rejection: study protocol of a randomized controlled pilot trial. Trials. 2019 Jan 11;20(1):37. doi: 10.1186/s13063-018-3158-6. PMID 30635033
- See also: Vienna Transplant and Complement Laboratory (VIETAC) website — http://www.vietac.at
- See also: Vitaeris website — http://www.vitaerisbio.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03444103/Prot_SAP_000.pdf